CLINICAL TRIAL: NCT04074382
Title: Functional Outcomes In Trauma Study - A Combined Retrospective and Prospective Cohort Study to Investigate Functional Outcomes Following Major Trauma.
Brief Title: FIT Study (Functional Outcomes In Trauma Study)
Status: Active, not recruiting | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: OR19/123401; 257064 (Other: IRAS Project ID (Health Research Authority, UK)); 19/YH/0280 (Other: Research Ethics Committee (REC) Reference)
Record Dates: First submitted 2019-08-27; First posted 2019-08-30 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2019-08

CONDITIONS: Patient Reported Outcome Measures; Recovery of Function; Rehabilitation; Disability Evaluation; Trauma Centers; Trauma Severity Indices; Advanced Trauma Life Support Care; Multiple Trauma/Injuries; Wounds and Injuries; Orthopedic Disorder; Surgery
Keywords: Patient Reported Outcome Measures; Recovery of Function; Rehabilitation; Disability Evaluation; Trauma Centers; Trauma Severity Indices; Advanced Trauma Life Support Care; Multiple Trauma/Injuries; Wounds and Injuries; Orthopedic Disorder; Surgery
MeSH Terms: conditions — Multiple Trauma; Wounds and Injuries; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Cohort: Prospective cohort (Phase 1, and Phase 2 Group A: explained in detailed description earlier) We will recruit and consent patients on the ward in the first few weeks following their admission for major trauma when the consultant in charge of their care feels that they are physically and emotionally/mentally ready and appropriate to take part in the study. A member of the research team will ask whether they want to take part in the study and offer them the participant information sheet. If happy to take part, the patient will have an account set up on the online questionnaire service we will be using called QTool. The consent form will be completed online at baseline along with the initial baseline PROM questionnaires. This group of people will then be sent reminders at 3, 6, 9 and 12 months to complete follow-up questionnaires, up to 28 days before or after these timepoints. They will then enter Phase 2 (Group A).
  Interventions: Other: Online Questionnaires; Other: Qualitative Interviews
- Retrospective Cohort: Retrospective cohort (Phase 1/2):
  Patients between 1 to 10 years following their major trauma will be identified using a database. We will randomly select which of these patients to include in our study, using computer software, to reduce selection bias, and those selected will be sent a recruitment pack in the post. We have calculated that we need at least 320 patients in the retrospective cohort to show any important changes.
  This group of patients will only complete the questionnaires once in phase 1, and once per year up to 10 years after their trauma in phase 2 (Group B).
  Interventions: Other: Online Questionnaires; Other: Qualitative Interviews

INTERVENTIONS:
Other: Online Questionnaires — We will use online questionnaires to complete research into functional outcomes after trauma
Other: Qualitative Interviews — We will undertake qualitative interviews (remote or face to face) to shed more light on reasons for functional outcomes after trauma

SUMMARY:
Why? There is not much information in the UK on how well patients who sustain major trauma function afterwards. Major trauma is defined as significant injuries with a calculated 'injury severity score' (ISS) over 15. The ISS is calculated based on how many parts of the body are injured and how badly injured these are, up to a maximum score of 75 (fatal). We feel that learning more about how these people cope afterwards, and what influences this will allow us to improve the care we can deliver in the future, which will hopefully lead to better outcomes.

What? We propose to implement the FIT (Functional outcomes In Trauma) study to assess how well patients function physically, psychologically and socially, and get back to activities of daily living, work and participation in recreational activities following major trauma.

Who? Major trauma patients: 2 cohorts: prospectively going forwards in time (from baseline to 12 months after trauma) and retrospectively going backwards in time (patients between 2-10 years after trauma).

Where? Leeds General Infirmary.

How? We will do this by collecting data from questionnaires completed by patients (also known as PROMS, or Patient Reported Outcome Measures), using an online questionnaire service developed at the University of Leeds, called QTool. These will offer the participants the chance to tell us how they are doing across lots of areas, with both tick-box multiple choice questions and open-ended questions to explain how they are doing and what influences this. We will also interview a random selection of patients in further detail to discuss how their trauma has affected them, how they found the study, how we could improve it. Afterwards we will send participants a copy of what we have learnt from the study and aim to publish it in a scientific journal.

Timeline/Phase overview:

The FIT Study will consist of 2 phases. Phase 1 will last for 2 years in total (12 months for prospective study cohort recruitment and 12 months follow-up for these patients) during which time data will be collected from the retrospective cohort as well.

Following this there will be a full analysis of the data, after which phase 2 of the FIT Study will begin.

Patients enrolled into phase 1 of the study will be given the option of consenting to being contacted annually to complete the same set of online PROMs, which will comprise phase 2 of the study. We will also continue active recruitment into both prospective and retrospective arms of the study in phase 2. We plan to continue data collection on an annual basis up to 10 years post trauma in phase 2 of the study for patients in both cohorts. We hope to incorporate elements of the FIT Study into future routine care with what we learn from the FIT Study, and develop our own unique Patient Reported Outcome Measure tool, with the overall aim of improving patient care and outcomes.

DETAILED DESCRIPTION:
Primary Research Questions/Objectives:

Research Questions:

1. How well do patients function physically following major trauma?
2. What influences this?
3. Which patient groups/injury patterns predict better outcome?
4. How long until a plateau of physical functioning is reached?

The primary aim of this project will be to assess the impact of major trauma, especially polytrauma (multiple body area trauma and injury) on the physical aspect of functional outcome (how well patients do physically after their trauma), the change over time and trends in this data, assessed by a questionnaire: the physical component score (PCS) of the Short Form-36 questionnaire, which will be our primary outcome measure. This is helps to assess how well people can physically function.

Physical function data will also be collected using other questionnaires including the the Trauma Outcomes Profile, Euroqol 5 Dimension Score, and Leeds Trauma Questionnaire, which will be secondary outcome measures.

Secondary Research Questions/Objectives:

Research Questions:

1. How well do patients function otherwise following major trauma, especially polytrauma (multiple body area injury)?
2. What influences this?
3. Which patient groups/injury patterns predict better outcome?
4. How long until a plateau of physical functioning is reached?
5. What are the unmet needs of the patient population?
6. How can we improve our service to meet the needs, and improve rehabilitation and functional outcomes after major trauma?

Secondary aims will include:

1. Assessing other areas of functional outcome (psychological wellbeing and mental function, social relations, and functional capacity) and quality of life of patients following discharge from hospital, and factors which affect this. This will be measured using 'patient reported outcome measures' questionnaires (PROMs) data, and the change in PROMs values in both prospective (going forward in time) and retrospective (going backwards in time) cohorts.
2. Assessing how trauma affects people's ability to work, which will be assessed using a targeted questionnaire as well as responses to the general questionnaires used.
3. How trauma affects patients' social, mobility, and care situation, which will be assessed using a targeted questionnaire.
4. Assessing the personal impact of trauma on the patient - how it has affected their lives most in various ways, and also assessing the changing needs of patients as they progress through their journey, their access to services, and opinions on how well the service we offer works for them. We will do this using a targeted qualitative questionnaire (open ended questions which lets them expand in their own words rather than just ticking yes/no/multiple choice answers). We will also include formal qualitative interviews (to a small group) with patients in person or over the phone/video link. This will allow for a powerful systematic analysis which will guide us to improve what we can offer to patients and reinforce the quality of care we deliver.
5. Assessing clinical progress following trauma, and how this relates to functional outcomes, using health records and imaging systems.
6. Feasibility study: We will also assess the feasibility of using similar questionnaires to assess functional outcomes, delivered in the same way as in the FIT Study, in usual care for patients at the Leeds Major Trauma Centre. This presents an exciting opportunity for a permanent positive change, and room for ongoing audit cycle, with a reliable mechanism for measurement.

Background and Rationale:

'Major trauma' is defined as patients having an accident so severe that it potentially poses an immediate threat to life, and depends on how many injuries a person sustains and their severity. The more injuries to more body areas a person sustains, the higher the threat to life. (1-5) Until recently, patients with multiple serious injuries (polytrauma) were not managed in the same way in all hospitals which led to unacceptably poor outcomes in certain cases. By 2013, across most of England, a major trauma network was set up to bring the most seriously injured patients to special 'major trauma centres' (MTCs) which are large hospitals with a lot of extra specialist teams available 24 hours a day, to respond to serious trauma. (5, 6) A recent report published evaluating the performance of the service developed highlighted significant improvements in both the care process and survival of patients after severe injury (7). Although we are saving more lives, in the UK we still lack longer term solid information on how well these patients function across all areas after discharge, in a way which can be measured and tracked.

'Functional outcome' has different components, and is broadly broken down into a person's physical functional ability, psychological wellbeing and mental function, social relationships with others, and ability to look after themselves and perform personal care and activities of daily living, work and engage with society as a whole. It can be measured on a scale according to how well a patient scores questionnaires designed to assess one of more of these areas, which have often been tested on large groups of people to work out what the average responses or scores would be for a given group. Changes to these scores can be tracked over time, and improvement or worsening of performance measured. Generally, these are referred to as Patient Reported Outcome Measures, or PROMs. (8, 9) We know from studies elsewhere, most notably Germany, that people's overall function (measured using PROMs) following serious injury can be affected for many years afterwards. (10-13) However, these are from countries with different populations, cultures and societies to the UK and in a different healthcare system. In the UK, other than one study which looked at 99 patients with moderate (45%) to severe (55%) injuries at 1-3 years after injury, there have been limited studies looking at functional outcomes in large numbers of major trauma patients. To the best of our knowledge, and when performing thorough literature review, there has been almost no published work done in the UK looking at functional outcome in patients with major trauma, including polytrauma, and none looking at this beyond 5 years. (14, 15)

We therefore intend to fill the knowledge gap in the UK on functional outcomes after major trauma, especially polytrauma, assessing functional outcomes using Patient Reported Outcome Measure forms (PROM's).

As we have managed a large number of patients with major trauma, including polytrauma, over the last 10 years, we have a large clinical database to use, as well as the large number of patients who will attend in the year ahead. In a relatively short time, we will be able to collect a lot of information on how patients function after major trauma from straight afterwards up to 10 years after their accident in a UK MTC setting, which should be relevant to other centres, and therefore useful information and potential learning points for the UK Trauma Network as a whole, which should benefit both hospitals and patients alike.

Hypotheses:

We hypothesise that physical function, as assessed by the Physical Component Score of the SF-36 PROM will continue to improve until 3 years, where we will see a significant difference in outcomes between groups, and then begin to plateau to a steadier level. We also hypothesise that the most rapid improvement will be in the first year following major trauma.

Null hypotheses:

The Physical Component Score of the SF-36 PROM will remain unchanged over time. Any change seen in the SF-36 physical component score will be the same across all timepoints.

Our hypotheses/null hypotheses are based on the limited literature which we have discussed in the background section, and also clinical experience which suggests that recovery is quickest in the first year, and by 2-3 years patients' physical function generally levels off. We hope to be able to determine which groups improve more than others and which factors affect this most, and show this on a graph over time, which will make the FIT study unique, and useful data to use in clinical practice. We also want to see if there are certain groups who do not follow this pattern and look into the reasons behind this.

Patient involvement in study design:

We arranged several focus group sessions to gather patient opinion on the various PROMS tools (numbers based, or quantitative responses), as well as the other more qualitative (more detailed, verbal response) questions which we wanted to explore. We incorporated the opinions of these patients into the design of the study, and also our Leeds Trauma Questionnaires which the patients had a lot of direct input to help design.

Methodology:

We felt that the best way to capture a meaningful set of information was to do set up a cohort study (looking at different groups at different points in time). In this way we could measure how well patients functioned who have already experienced major trauma, and especially polytrauma, (back in time, or retrospective cohort), and patients who experience major trauma right from the beginning of their journey and how their functional outcomes change over time going forwards (prospective cohort). We also wanted to include a feasibility study as part of the FIT Study, to see how patients/participants felt about the questionnaires used and whether we needed to improve anything, especially if we were to use the questionnaires in usual care rather than just as part of a research study in the future.

Questionnaires to be used:

1. Background questionnaire about patients' work, social, care and mobility circumstances (and how this was affected by their major trauma). Patients in the different cohorts will answer slightly different versions of this depending on whether they have completed sections of it before or not.
2. Euroqol 5 Dimensions score (EQ-5D): This offers a good short snapshot of how well a patient is doing, with five questions covering five broad areas and asks how well someone is feeling on a scale from 1-100. We can also calculate how much we need to spend to improve someone's quality of life using this questionnaire which will be interesting.
3. Short Form Health Survey 36 (SF-36): This is one of the most widely used PROMs, and looks at 8 areas of overall function, including physical function. We have chosen this as our main measurement because we know it is reliable and widely tested and is good at showing change over time so we can measure how well people improve in our study.
4. Trauma Outcomes Profile (TOP): This is a questionnaire designed specifically to look at people who have undergone trauma across a range of areas and allows people to give specific ratings about how much they are bothered by pain and limited function in different body areas. We have also included a few extra questions along with this which ask about sleep (from the Sleep Condition Indicator).
5. HADS (Hospital Anxiety and Depression Scale) - This is a questionnaire to assess mood, chosen because it is short and easy to complete, and doesn't include any questions about physical symptoms of depression which could be influenced by injuries from trauma.
6. Leeds Trauma Questionnaire - This is a free-space qualitative questionnaire we have designed. It asks patients to list which of their injuries bother them most and why, what their changing needs are over time, expectation of improvement, and about their time at our hospital and any areas they would like to see improve.

Retrospective cohort (Phase 1):

Patients between 1 to 10 years following their major trauma will be identified using a database. We will randomly select which of these patients to include in our study, using computer software, to reduce selection bias, and those selected will be sent a recruitment pack in the post. This will include an invite letter, participant information sheet, and details of how to log in to the online questionnaire service we will be using, called QTool, straight away if they wish and complete the questionnaires. We will also give them the opportunity of letting us know they do not wish to take part. We will allow patients at least 7 days to let us know they don't want to take part or to log into their online QTool account by themselves, and after this telephone them to see if they would be happy to take part or want more information before signing up. If we have not managed to speak with them by 14 days and they have not got in touch with us or signed up to the study, we will send them another letter. We will send up to a maximum of 4 letters to the patient to invite them to take part. We know from several other studies that there is a poor initial response rate of approximately 15%, but that with each subsequent round of invitations this increases by another 15% each time. We have calculated that we need at least 320 patients in the retrospective cohort to show any important changes, and also want to minimise recruitment bias - this is the main area of our study at risk of bias. If we persist in contacting patients in relatively small waves we will maximise recruitment of a larger proportion of patients who have been identified as eligible, and therefore get a more accurate picture of overall functional outcomes in these patients. This group of patients will only complete the questionnaires once in phase 1, and once per year up to 10 years after their trauma in phase 2 (Group B).

Prospective cohort (Phase 1, and Phase 2 Group A: explained below) We will recruit and consent patients on the ward in the first few weeks following their admission for major trauma when the consultant in charge of their care feels that they are physically and emotionally/mentally ready and appropriate to take part in the study. A member of the research team will ask whether they want to take part in the study and offer them the participant information sheet. If happy to take part, the patient will have an account set up on the online questionnaire service we will be using called QTool. The consent form will be completed online at baseline along with the initial baseline PROM questionnaires. This group of people will then be sent reminders at 3, 6, 9 and 12 months to complete follow-up questionnaires, up to 28 days before or after these timepoints. They will then enter phase 2 (Group A) as described below.

Phase 1 recruitment will take place from 1 September 2019 with active recruitment until September 2020. The patients in the prospective cohort will be followed up for 12 months, with the final patient completing their 12 month follow-up questionnaire by September 2021. During this time, retrospective participants will also be recruited.

All cohorts and groups:

Patients will be able to complete their online questionnaires wherever they feel most comfortable. When an inpatient we will provide a computer for the prospective group to use. We will also provide a computer for either group to use in the hospital once discharged if they do not have access to one at home, or if they would prefer to complete it at any orthopaedic outpatient follow-up clinic appointment they have at the hospital.

We will also collect information from our clinical systems about the patients' medical conditions and how well their injuries heal/healed as they progress through their journey. We can then link the PROMs scores to their medical conditions and injuries and which affect functional outcome most. We will also collect information about where they live and see if this also affects how well they do afterwards.

Qualitative interviews (Phase 1):

5 to 10 patients from each cohort will be invited to an interview (either in person at the hospital or over the phone or video link) to discuss their feelings about all areas of the study, and also to ask them about their injuries and how they have affected them in detail, which aspects affected them most, what their main needs are and how they have changed, what advice they would give to others in their situation, and feedback on their experience at our centre; we will use the Leeds Trauma Questionnaire as a basis for this part of the interview. The interview process will be supervised by an experienced psychologist to ensure that any bias in how the questions in the interviews are posed is kept to a minimum.

Phase 2:

After the first part of the study (phase 1) we will analyse the information we have collected, and then go ahead with the second phase. All patients who were part of phase 1 will automatically be included (and will have consented for this), and we will also recruit more people into the prospective cohort of the study. Participants in phase 2 will answer questionnaires up until 10 years following their major trauma.

To summarise, there will be 2 groups of patients, A and B:

Group A will be patients new to the FIT Study, recruited in the same way as for phase 1, but only prospectively (going forwards in time). These will be patients who were not previously involved in phase 1. They will complete the same sets of questionnaires as those in phase 1 did. Once they have completed the same set of questions as those participants in phase 1, they will move into group B.

Group B will be patients who have already completed either phase 1 of the FIT study (and consented to take part in phase 2), or have come from Group A of Phase 2. Participants who have already been in the study will be given the same standard PROMs to answer as before, but the Leeds Trauma Questionnaire will be slightly different for them so we don't repeat questions we already know the answers to.

Phase 2 recruitment of new patients will begin on 1 January 2021, and finish on 1 January 2029; it will finish on 1 January 2031 after the final patient in Group A (recruited in 2029) has finished their 12 month questionnaire follow-up.

Analysis:

Our aim is to analyse the data in a way that we should be able to predict how patients will do at 2-3 years based on their initial medical problems and injuries, and discover what other aspects are important at predicting outcome. We aim to link replies to the open-ended words based (qualitative) questionnaires and interviews with the numbersbased (quantitative) tick-box based PROMs, to hopefully help give further depth and explanation into reasons behind different people's scores.

1. Descriptive statistics:

   In general, summary statistics [n (number of available measurements; arithmetic mean, standard deviation, median, minimum and maximum] for quantitative variables and absolute and relative frequency tables for qualitative data will be presented. We will summarise using descriptive statistics for key timepoints following trauma.
2. Analytical model of quantitative data:

   We will be using a sophisticated mixed effects "latent class" regression model, which should facilitate predictive growth modelling. This is a model which allows us to group subjects into different classes or types, whose phenotype can plotted into different outcome trajectories against time. These classes or types can be made up of individual or clustered subgroups. We anticipate 3 types of outcome trajectories for our cohort. This should allow us to predict functional outcome based on patient and injury characteristics and increase the utility of our study.
3. Analysis of Qualitative data:

   We will perform a thematic analysis, using NVivo software. We will use a systematic approach to familiarisation, identification and indexing of key themes, and viewing these in the context of the quantitative PROMS score changes.

   We will present these results descriptively.
4. Synthesis We will aim to synthesise quantitative and qualitative data in our analysis, in order to correlate and provide a contextual framework to help assess quantitative data along with narrative data.

Publication:

We will aim to publish our study in a high profile scientific journal, and will distribute a summary of our study findings to all participants after phase 1, and throughout and at the end of phase 2.

References:

1. Balogh ZJ, Varga E, Tomka J, Suveges G, Toth L, Simonka JA. The new injury severity score is a better predictor of extended hospitalization and intensive care unit admission than the injury severity score in patients with multiple orthopaedic injuries. Journal of Orthopaedic Trauma. 2003;17(7):508-12. PubMed PMID: 12902789.
2. Abajas Bustillo R, Amo Setien FJ, Ortego Mate MDC, Segui Gomez M, Dura Ros MJ, Leal Costa C. Predictive capability of the injury severity score versus the new injury severity score in the categorization of the severity of trauma patients: a cross-sectional observational study. European Journal of Trauma & Emergency Surgery. 2018;08:08. doi: https://dx.doi.org/10.1007/s00068-018-1057-x. PubMed PMID: 30535521.
3. Boyd CR, Tolson MA, Copes WS. Evaluating trauma care: the TRISS method. Trauma Score and the Injury Severity Score. Journal of Trauma-Injury Infection & Critical Care. 1987;27(4):370-8. PubMed PMID: 3106646.
4. Palmer C. Major trauma and the injury severity score--where should we set the bar? Annual proceedings / Association for the Advancement of Automotive Medicine Association for the Advancement of Automotive Medicine.

   2007;51(pp 13-29). PubMed PMID: 352407356.
5. NCEPOD:, Findlay G, Martin I, Carter S, Smith N, Weyman D, et al. Trauma: Who cares? A report of the National Confidential Enquiry into Patient Outcome and Death (2007). 4-8 Maple Street, London W1T 5HD: Published November 2007 by the National Confidential Enquiryinto Patient Outcome and Death (2007), 2007 Contract No.: ISBN 0-9539240-8-4.
6. Morse A, Fisher A, Ross C, Henderson C, Kirk S, Feroze M, et al. Major trauma care in England: National Audit Office Report. National Audit Office Press Office 157-197 Buckingham Palace Road Victoria LondonSW1W 9SP: National Audit Office, 2010.
7. Moran C, Lecky F, Bouamra O, Lawrence T, Edwards A, Woodford M, et al. Changing the System - Major Trauma

   Patients and Their Outcomes in theNHS (England) 2008-17. EClinicalMedicine, The Lancet [Internet]. 2018; (2-3 ):

   [13-21 pp.]. Available from: https://www.thelancet.com/action/showPdf?pii=S2589-5370%2818%2930 007-5.
8. Pirente N, Ottlik Y, Lefering R, Bouillon B, Neugebauer E, Grimme K, et al. Quality of life in multiply injured patients:

   Development of the Trauma Outcome Profile (TOP) as part of the modular Polytrauma Outcome (POLO) Chart.

   European Journal of Trauma. 2006;32(1):44-62. doi: http://dx.doi.org/10.1007/s00068-006-0150-8. PubMed PMID:

   43428261.
9. McDowell I. Measuring Health: A Guide to Rating Scales and Questionnaires. Third Edition ed. Oxford, UK: Oxford University Press; 2006. 765 p.
10. Zwingmann J, Hagelschuer P, Langenmair E, Bode G, Herget G, Sudkamp NP, et al. Lower health-related quality of life in polytrauma patients long-term follow-up after over 5 years. Medicine. 2016;95(19). doi: http://dx.doi.org/10.1097/MD.0000000000003515. PubMed PMID: 610532475.
11. Falkenberg L, Zeckey C, Mommsen P, Winkelmann M, Zelle BA, Panzica M, et al. Long-term outcome in 324 polytrauma patients: What factors are associated with posttraumatic stress disorder and depressive disorder symptoms? European Journal of Medical Research. 2017;22(1). doi: http://dx.doi.org/10.1186/s40001-017-0282-9.

    PubMed PMID: 618987349.
12. Zeckey C, Hildebrand F, Pape HC, Mommsen P, Panzica M, Zelle BA, et al. Head injury in polytrauma-Is there an effect on outcome more than 10 years after the injury? Brain Injury. 2011;25(6):551-9. doi: http://dx.doi.org/10.3109/02699052.2011.568036. PubMed PMID: 361697849.
13. Attenberger C, Amsler F, Gross T. Clinical evaluation of the Trauma Outcome Profile (TOP) in the longer-term follow-up of polytrauma patients. Injury. 2012;43(9):1566-74. doi: http://dx.doi.org/10.1016/j.injury.2011.01.002. PubMed PMID: 51238702.
14. Spreadborough S, Radford K, das Nair R, Brooks A, Duffy M. A study of outcomes of patients treated at a UK major trauma centre for moderate or severe injuries one to three years after injury. Clinical rehabilitation. 2018;32(3):410-8.

    doi: http://dx.doi.org/10.1177/0269215517730862. PubMed PMID: 623852730.
15. Folkard SS, Bloomfield TD, Page PRJ, Wilson D, Ricketts DM, Rogers BA. Factors affecting planned return to work after trauma: A prospective descriptive qualitative and quantitative study. Injury. 2016;47(12):2664-70. doi: http://dx.doi.org/10.1016/j.injury.2016.09.040. PubMed PMID: 613549820.

ELIGIBILITY:
Inclusion Criteria:

* Injury Severity Score >15
* Age 18-65

Exclusion Criteria:

* Impaired capacity of patient or proxy (dementia, significantly reduced cognitive ability)
* Patient not deemed to be in a physical or mental state to provide consent
* Any isolated head injury
* Involvement in another study, and these would adversely impact one another
* No access to internet linked device to complete questionnaires
* Poor grasp of English language
* Patient deceased

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated at Leeds Teaching Hospitals, who sustained/sustain major trauma (with priority for inclusion given to polytrauma) - to assess functional outcomes in these patients
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2031-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Physical Component Score of SF-36v2 - PROM | As per description: 0-10 years after trauma. We will aim to collect this data in phase 1 and phase 2.
  The primary aim of this project will be to assess the impact of major trauma, especially polytrauma, on the physical aspect of functional outcome, the change over time and trends in this data, assessed by the physical component score (PCS) of the SF-36 as our primary outcome measure.
  The SF-36 is a 36 item form, developed in 1990 based on work from the Rand corporation's Medical Outcomes Study in the 1970's is a widely used and validated measure of general function, covering eight domains (physical functioning, role limitations due to physical and emotional problems, bodily pain, social functioning, general mental health, vitality, general health perceptions). It has been extensively validated globally, and used in a large number of functional outcome studies which will allow broad comparison with our study group. We will use the Physical Component Score as our primary outcome measure

SECONDARY OUTCOMES:
Trauma and Outcomes Profile (TOP) - PROM | As per description: 0-10 years after trauma. We will aim to collect this data in phase 1 and phase 2.
  This is a questionnaire designed specifically to look at people who have undergone trauma across a range of areas and allows people to give specific ratings about how much they are bothered by pain and limited function in different body areas. We have also included a few extra questions along with this which ask about sleep (from the Sleep Condition Indicator).
HADS: Hospital Anxiety and Depression Score - PROM | As per description: 0-10 years after trauma. We will aim to collect this data in phase 1 and phase 2.
  This is a 14 item form, designed by Prof Snaith (Leeds, UK) in 1983, specifically to measure non-physical symptoms of anxiety and depression. It is a widely used and validated questionnaire. It is most useful in cases where there may be other reasons to explain physical aspects of depression, which may include change to appetite and sleep for example; trauma patients may experience many of the same symptoms but due to pain and injury rather than depression/anxiety. We therefore feel that this would be the most appropriate scale to use to measure the effect of trauma on mental health. It is also short, to reduce question burden.
EQ-5D: Euroqol 5 Dimensions Scale | As per description: 0-10 years after trauma. We will aim to collect this data in phase 1 and phase 2.
  This is a 5-item short form comprising of five questions covering five broad domains (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) as well as a visual analogue rating scale (VAS) of overall health status. It is quick to complete, and provides a good snapshot of function, and also allows for calculation of Quality Adjusted Life Years (QALYs) to assess the relative economic benefit of interventions. It is a widely used and validated instrument, and also allows for comparison to other population and study groups.
Leeds Trauma Questionnaire - PROM/PREM | As per description: 0-10 years after trauma. We will aim to collect this data in phase 1 and phase 2.
  The Leeds Trauma Questionnaire is a selection of closed and open-ended questions to obtain useful quantitative and qualitative data, primarily focussing on the personal impact of trauma on the patients, how their needs have changed over time, and an element of service evaluation and areas for improvement - serving as a Patient Reported Experience Measure (PREM), with one question also focussing on self-efficacy. We have called this the "Leeds Trauma Questionnaire", and it will vary depending on the timepoint the questions are being asked, hence reference to versions 1-4 in the prospective cohort (phase 1, and phase 2 group A), and version 5 for phase 2 Group B. Version 5 will be almost identical to version 4. The retrospective cohort (phase 1) will complete all parts of this.
Qualitative Interview Outcomes | As per description: 0-10 years after trauma. We will aim to collect this data in phase 1.
  5-10 patients from each cohort will be invited to take part in an interview for a combined feasibility study and discussion about their experience:
  1. To ascertain which of the questionnaires were most useful to them and how easy they were to complete. We will also ask if they feel there are any areas which should be addressed which have not been.
  2. To assess the personal impact of trauma on the patient - how it has affected their lives most in various ways, and also assessing the changing needs of patients as they progress through their journey, their access to services, and opinions on how well the service we offer works for them.

OTHER OUTCOMES:
Work Status | As per description: 0-10 years after trauma. We will aim to collect this data in phase 1 and phase 2.
  2) Assessing how trauma affects people's ability to work, which will be assessed using a targeted questionnaire as well as responses to the general questionnaires used.
Social and Care Status | As per description: 0-10 years after trauma. We will aim to collect this data in phase 1 and phase 2.
  3) How trauma affects patients' social, mobility, and care situation, which will be assessed using a targeted questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Peter Giannoudis, MD, Study Chair — Leeds Teaching Hospitals; Paul Andrzejowski, BMBS, Principal Investigator — Leeds Teaching Hospitals
Locations (1):
- Leeds teaching Hospitals, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
As part of the participant information sheet and consent form, it will be made clear to patients that taking part in the study will require suitably authorised members of the research team to view their medical records, and that their information gathered from the records and from the study may also be used for future research or, once anonymised, shared with other researchers. The patient must consent to all elements of this in order to take part in the study, and their wishes not to take part will be respected. We have no current defined plans for data sharing, but may do so with suitable teams in the future.

REFERENCES:
- [Background] Balogh ZJ, Varga E, Tomka J, Suveges G, Toth L, Simonka JA. The new injury severity score is a better predictor of extended hospitalization and intensive care unit admission than the injury severity score in patients with multiple orthopaedic injuries. J Orthop Trauma. 2003 Aug;17(7):508-12. doi: 10.1097/00005131-200308000-00006. PMID 12902789
- [Background] Abajas Bustillo R, Amo Setien FJ, Ortego Mate MDC, Segui Gomez M, Dura Ros MJ, Leal Costa C. Predictive capability of the injury severity score versus the new injury severity score in the categorization of the severity of trauma patients: a cross-sectional observational study. Eur J Trauma Emerg Surg. 2020 Aug;46(4):903-911. doi: 10.1007/s00068-018-1057-x. Epub 2018 Dec 8. PMID 30535521
- [Background] Boyd CR, Tolson MA, Copes WS. Evaluating trauma care: the TRISS method. Trauma Score and the Injury Severity Score. J Trauma. 1987 Apr;27(4):370-8. PMID 3106646
- [Background] Palmer C. Major trauma and the injury severity score--where should we set the bar? Annu Proc Assoc Adv Automot Med. 2007;51:13-29. PMID 18184482
- [Background] Moran CG, Lecky F, Bouamra O, Lawrence T, Edwards A, Woodford M, Willett K, Coats TJ. Changing the System - Major Trauma Patients and Their Outcomes in the NHS (England) 2008-17. EClinicalMedicine. 2018 Aug 5;2-3:13-21. doi: 10.1016/j.eclinm.2018.07.001. eCollection 2018 Aug-Sep. PMID 31193723
- [Background] Lefering R, Tecic T, Schmidt Y, Pirente N, Bouillon B, Neugebauer E; POLO Chart Study Group. Quality of life after multiple trauma: validation and population norm of the Polytrauma Outcome (POLO) chart. Eur J Trauma Emerg Surg. 2012 Aug;38(4):403-15. doi: 10.1007/s00068-011-0149-7. Epub 2011 Sep 14. PMID 26816121
- [Background] Zwingmann J, Hagelschuer P, Langenmair E, Bode G, Herget G, Sudkamp NP, Hammer T. Lower Health-Related Quality of Life in Polytrauma Patients: Long-Term Follow-Up After Over 5 Years. Medicine (Baltimore). 2016 May;95(19):e3515. doi: 10.1097/MD.0000000000003515. PMID 27175646
- [Background] Falkenberg L, Zeckey C, Mommsen P, Winkelmann M, Zelle BA, Panzica M, Pape HC, Krettek C, Probst C. Long-term outcome in 324 polytrauma patients: what factors are associated with posttraumatic stress disorder and depressive disorder symptoms? Eur J Med Res. 2017 Oct 30;22(1):44. doi: 10.1186/s40001-017-0282-9. PMID 29084612
- [Background] Zeckey C, Hildebrand F, Pape HC, Mommsen P, Panzica M, Zelle BA, Sittaro NA, Lohse R, Krettek C, Probst C. Head injury in polytrauma-Is there an effect on outcome more than 10 years after the injury? Brain Inj. 2011;25(6):551-9. doi: 10.3109/02699052.2011.568036. PMID 21534733
- [Background] Attenberger C, Amsler F, Gross T. Clinical evaluation of the Trauma Outcome Profile (TOP) in the longer-term follow-up of polytrauma patients. Injury. 2012 Sep;43(9):1566-74. doi: 10.1016/j.injury.2011.01.002. Epub 2011 Jan 20. PMID 21255778
- [Background] Spreadborough S, Radford K, das Nair R, Brooks A, Duffy M. A study of outcomes of patients treated at a UK major trauma centre for moderate or severe injuries one to three years after injury. Clin Rehabil. 2018 Mar;32(3):410-418. doi: 10.1177/0269215517730862. Epub 2017 Sep 20. PMID 28929802
- [Background] Folkard SS, Bloomfield TD, Page PRJ, Wilson D, Ricketts DM, Rogers BA. Factors affecting planned return to work after trauma: A prospective descriptive qualitative and quantitative study. Injury. 2016 Dec;47(12):2664-2670. doi: 10.1016/j.injury.2016.09.040. Epub 2016 Sep 30. PMID 27712904